CLINICAL TRIAL: NCT05636267
Title: A Multicenter, Open-Label, Phase Ib/II Study of AK119 and AK112 With or Without Chemotherapy in Patients With EGFR-mutant Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Who Have Failed to Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) Treatment
Brief Title: Study of AK119 and AK112 With or Without Chemotherapy for NSCLC Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK119-201
Record Dates: First submitted 2022-11-09; First posted 2022-12-05 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AK119 + AK112 (Experimental): Subjects will receive AK119 plus AK112 via intravenously (IV) Q3W, up to 2 years.
  Interventions: Drug: AK119; Drug: AK112
- AK119 + AK112 + Pemetrexed + Carboplatin (Experimental): Subjects will receive AK119 and AK112 plus pemetrexed and carboplatin via intravenously (IV) Q3W, up to 4 cycles. Afterward, AK119 and AK112 plus pemetrexed will continue to be treated up to 2 years.
  Interventions: Drug: AK119; Drug: AK112; Drug: Pemetrexed; Drug: Carboplatin
- AK112 (Experimental): Subjects will receive AK112 monotherapy via intravenously (IV) Q3W, up to 2 years.
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK119 — AK119 IV every 3 weeks.
  Arms: AK119 + AK112; AK119 + AK112 + Pemetrexed + Carboplatin
Drug: AK112 — AK112 IV every 3 weeks.
Drug: Pemetrexed — Pemetrexed IV every 3 weeks.
  Arms: AK119 + AK112 + Pemetrexed + Carboplatin
Drug: Carboplatin — Carboplatin IV every 3 weeks.
  Arms: AK119 + AK112 + Pemetrexed + Carboplatin

SUMMARY:
This is a phase Ib/II study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of AK119 and AK112 With or Without Chemotherapy for NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and voluntarily sign the written informed consent, which must be signed before the designated research procedure.
2. Age ≥ 18 and ≤ 75, male or female.
3. Local advanced or metastatic non-squamous NSCLC confirmed by histology or cytology according to eighth edition of the TNM classification for lung cancer.
4. EGFR activating mutation confirmed by tumor histology, cytology or hematology.
5. Failed to previous EGFR-TKI treatment.
6. ECOG performance status 0 to1.
7. Life expectancy ≥3 months.
8. At least one measurable lesion according to RECIST v1.1.
9. Adequate organ function.

Exclusion Criteria:

1. Histological or cytological pathology confirmed the presence of small cell carcinoma or squamous cell carcinoma.
2. Have suffered from the second primary active malignant tumor in the past 3 years.
3. There are other driving gene mutations that can obtain effective treatment.
4. Receipt of the following treatments or procedures: immunotherapy, including immunocheckpoint inhibitors, immunocheckpoint agonists, immunocellular therapy, and any other treatment targeting tumor immune mechanism; systematic chemotherapy in the advanced stage (IIIB-IV); anti-angiogenesis drugs, except for small molecule anti-angiogenesis drugs with drug withdrawal more than 4 weeks; extensive radiotherapy within 4 weeks; EGFR-TKIs within 2 weeks.
5. Symptomatic central nervous system metastases.
6. The toxicity of previous anti-tumor therapy has not been alleviated.
7. Uncontrolled massive ascites, pleural effusion or pericardial effusion.
8. Active autoimmune diseases in the past 2 years.
9. History of interstitial lung disease or noninfectious pneumonitis.
10. Suffering from clinically significant cardiovascular or cerebrovascular diseases.
11. History of severe bleeding tendency or coagulation dysfunction.
12. History of deep vein thrombosis, pulmonary embolism or any other serious thromboembolism in the past 3 months.
13. Serious infection in the past 4 weeks.
14. Acute exacerbation of chronic obstructive pulmonary disease or asthma in the past 4 weeks.
15. History of human immunodeficiency virus (HIV) infection.
16. History of severe hypersensitivity reactions to other mAbs.
17. History of organ transplantation.
18. Any other conditions that, in the opinion of the investigator, may increase the risk when receiving the investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | During the first 3 weeks
  DLTs will be assessed during the first 3 weeks of treatment. DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT observation period.
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST Version 1.1).
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST Version 1.1).
Duration of response (DoR) | Up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to 2 years
  TTR is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR (based on RECIST Version 1.1).
Overall survival (OS) | Up to 2 years
  OS defined as the time from the first dose to death from any cause.
Maximum observed concentration (Cmax) of AK119 and AK112 | From first dose of study drug through last dose
  The PK parameters include serum concentrations of AK119 and AK112 at different timepoints after study drug administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through last dose
  The immunogenicity of AK119 and AK112 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, China